CLINICAL TRIAL: NCT01369875
Title: Phase II Study of Lymphocytes Generated With Engineered Cells for Costimulation Enhancement in Patients With Metastatic Melanoma Following Lymphodepletion
Brief Title: Modified Tumor Infiltrating Lymphocytes for Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature closure. Protocol did not meet its primary objective.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110163; 11-C-0163
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Immunotherapy; Cell Therapy; Metastatic Cancer; Melanoma; Metastatic Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasm Metastasis | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Young TIL (Experimental): Tumor Infiltrating Lymphocytes : intravenous (IV) over 30 minutes on day 0
  Aldesleukin : 720,000 IU/kg IV over 15 min every 8 hours (+/- 1hr) beginning within 24 hours of cell infusion and continuing for up to 5 days (max. 15 doses.)
  Fludarabine : 25 mg/m2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days (days -5 to -1)
  Cyclophosphamide : 60 mg/kg/day X 2 days IV over 1 hour on days -7 and -6
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Aldesleukin; Biological: Tumor Infiltrating Lymphocytes
- ECCE Young TIL (Experimental): Tumor Infiltrating Lymphocytes : IV over 30 minutes on day 0
  Aldesleukin : 720,000 IU/kg IV over 15 min every 8 hours (+/- 1hr) beginning within 24 hours of cell infusion and continuing for up to 5 days (max. 15 doses.)
  Fludarabine : 25 mg/m2/day IVPB daily over 30 minutes for 5 days (days -5 to -1)
  Cyclophosphamide : 60 mg/kg/day X 2 days IV over 1 hour on days -7 and -6
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Aldesleukin; Biological: Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Drug: Cyclophosphamide — 60 mg/kg/day X 2 days intravenous (IV) over 1 hour on days -7 and -6
  Other Names: Cytoxan
Drug: Fludarabine — 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days (days -5 to -1)
  Other Names: Fludara
Biological: Aldesleukin — 720,000 IU/kg intravenous (IV) over 15 min every 8 hours (+/- 1hr) beginning within 24 hours of cell infusion and continuing for up to 5 days (max. 15 doses.)
  Other Names: IL-2
Biological: Tumor Infiltrating Lymphocytes — Intravenous (IV) over 30 minutes on day 0

SUMMARY:
Background:

- Tumor infiltrating lymphocytes (TIL) are white blood cells that have been taken from tumor tissue. The cells are modified to help them kill tumor cells, then given back to the person with cancer. By giving these cells to patients, researchers hope to improve the current treatments available for patients with melanoma that has not responded to standard therapies. The TIL will be given after treatments that will suppress the immune system. This makes it easier for the TIL to attack the cancer cells. The TIL will also be given with aldesleukin (IL-2), which is designed to help keep the TIL cells alive in the body.

Objectives:

- To study the safety and effectiveness of specially modified tumor infiltrating lymphocytes to treat melanoma that has not responded to other treatments.

Eligibility:

- Individuals at least 18 years of age who have metastatic melanoma that has not responded to other treatments.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood tests and imaging studies.
* A piece of tumor will be collected and white blood cells will be separated to make the TIL for the treatment.
* Participants will take drugs to suppress the immune system for 7 days before the start of treatment.
* Participants will receive the TIL in a single dose. Then they will receive IL-2 every 8 hours for up to 15 doses. Participants will remain in the hospital for up to 2 weeks after treatment. They will be monitored with frequent blood tests and other studies.
* After leaving the hospital, participants will have regular followup visits every 1 to 4 months for the first year. Then they will return for followup every 3 to 4 months, as directed by the study researchers.

DETAILED DESCRIPTION:
Background:

* Tumor Infiltrating Lymphocyte (TIL) administration and high dose interleukin (IL)-2 following lymphodepletion can mediate durable complete responses in patients with refractory melanoma. Obstacles to administration of this therapy include failure to establish TIL in vitro for about 20% of patients, long delays between tumor resection and TIL establishment resulting in poor TIL attributes for therapy and patient ineligibility due to progression, and requirements for large numbers of feeder cells for TIL expansion to therapeutic numbers.
* The K562 cell line was engineered to express the 4-1BBL costimulatory molecule and CD64 (the high affinity Fc receptor for loading with antibodies such as OKT3). The K562.CD64.4-1BBL Engineered Cells with Costimulation Enhancement (ECCE) replaced up to 75% of feeder cells in large scale TIL expansions. ECCE added to tumor cell suspensions provided costimulation in trans resulting in rapid and reliable lymphocyte growth even from tumors with no TIL growth under standard conditions.
* A cloned K562.CD64.4-1BBL-7F11 ECCE line was produced under Good Manufacturing Practice (GMP) conditions and a master cell bank has been generated. An optimized protocol was established to rapidly expand (REP) young TIL using minimum feeders and 7F11. These ECCE REPed TIL retained tumor recognition and some other attributes of standard TIL, but differed from standard TIL by containing fewer CD4+ cells and more natural killer cells.

When 7F11ECCE were added directly to single cell tumor suspensions, young TIL cultures were reliably generated even from patients who otherwise would not have a standard young TIL culture for treatment.

Objectives:

Primary objectives:

* In cohort 1, to evaluate whether young TIL that are rapidly expanded using 7F11 ECCE to replace some feeder cells and administered with IL-2 in patients following a non -myeloablative conditioning regimen will result in clinical tumor regression in patients with refractory metastatic melanoma.
* In Cohort 2, to evaluate whether young TIL generated using in trans costimulation with 7F11 ECCE in patients for whom standard young TIL did not grow can mediate tumor regression after a nonmyeloablative conditioning with high dose IL-2 in patients with refractory metastatic melanoma.
* Determine the toxicity of ECCE young TIL in these treatment regimens

Eligibility:

Patients who are 18 years of age or older must have:

* metastatic melanoma;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* One or more lesions 2 cm or greater suitable for resection for TIL culture

Patients may not have:

* Concurrent major medical illnesses;
* Any form of immunodeficiency;
* Severe hypersensitivity to any of the agents used in this study;
* Contraindications for high dose IL-2 administration.

Design:

* Patients will undergo resection to obtain tumor for generation of autologous young TIL cultures.
* Parallel TIL cultures will be established using a) the standard technique with IL-2 only and b) the Engineered Cells with Costimulation Enhancement (ECCE) protocol using irradiated K562.CD64.4-1BBL-7F11 (7F11) cells.
* After 10 to 20 days cultures will undergo evaluation for TIL establishment. Standard TIL will be used preferentially and patients who have TIL established by standard methods will be assigned to Cohort 1
* Cohort 1:

  * TIL will undergo ECCE REP by exposure to OKT-3, IL-2, feeder cells and irradiated 7F11.
  * Patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day intravenous (IV)) on days -7 and -6 and fludarabine (25 mg/m^2/day IV) on days -5 through -1.
  * On day 0 patients will receive the infusion of autologous young TIL and then begin highdose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).
  * Clinical and immunologic response will be evaluated about 4-6 weeks after treatment.
  * Using an optimal two-stage Phase II design, initially 18 patients will be enrolled, and if three or more of the first 18 patients have a clinical response (partial response (PR) or complete response (CR)), accrual will continue to 35 patients, targeting a 30% goal for objective response.
* If standard young TIL fail to grow then ECCE young TIL will be evaluated and patients who have ECCE TIL available will be assigned to Cohort 2 .
* Cohort 2:

  * Cultures from patients in Cohort 2 will be evaluated for ECCE TIL establishment. If adequate ECCE TIL are available, TIL will undergo ECCE REP by exposure to OKT-3, IL-2, feeder cells and irradiated 7F11.
  * Patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m^2/day IV) on days -5 through -1.
  * On day 0 patients will receive the infusion of autologous young TIL and then begin highdose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).
  * Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion.
  * Using a small optimal two-stage Phase II design, initially 9 patients will be enrolled, and if one or more of the first 9 patients has a clinical response (PR or CR), accrual will continue to 24 patients, targeting a 25% goal for objective response.
* If TIL cultures were not established by either standard methods or ECCE young TIL protocols, patients will be eligible for re-resection and evaluation of TIL from a different site.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic melanoma with at least one lesion that is resectable for tumor infiltrating lymphocytes (TIL) generation.
  2. Patients with 3 or less brain metastases are eligible. Note: If lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
  3. Greater than or equal to 18 years of age.
  4. Willing to sign a durable power of attorney
  5. Able to understand and sign the Informed Consent Document
  6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  7. Life expectancy of greater than three months.
  8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
  9. Serology:

     1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients engineered cells with costimulation enhancement (ECCE) TIL 14 who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     2. Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
     3. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
  10. Hematology:

      1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
      2. White blood cell (WBC) (> 3000/mm^3).
      3. Platelet count greater than 100,000/mm^3.
      4. Hemoglobin greater than 8.0 g/dl.
  11. Chemistry:

      1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  12. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
  13. Six weeks must have elapsed since any prior anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy to allow antibody levels to decline.
  14. Patients who have previously received any anti-CTLA4 antibody and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Systemic steroid therapy required.
3. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who ECCE TIL 15 have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms
8. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
9. Documented LVEF of less than or equal to 45% tested in patients with:

   * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   * Age greater than or equal to 60 years old
10. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking
    * Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2012-02-13 (Actual); Study Completion 2012-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Atkins MB, Lotze MT, Dutcher JP, Fisher RI, Weiss G, Margolin K, Abrams J, Sznol M, Parkinson D, Hawkins M, Paradise C, Kunkel L, Rosenberg SA. High-dose recombinant interleukin 2 therapy for patients with metastatic melanoma: analysis of 270 patients treated between 1985 and 1993. J Clin Oncol. 1999 Jul;17(7):2105-16. doi: 10.1200/JCO.1999.17.7.2105. PMID 10561265
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0163.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Young TIL | ECCE Young TIL
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Young TIL | ECCE Young TIL | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 | 46.0 | 48.0 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Tumor Regression.
Description: Clinical tumor regression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progression (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD.
Time Frame: up to approximately 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Young TIL | ECCE Young TIL
Number analyzed (Participants) | 1 | 1
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Progression | 1 | 1
  Stable Disease | 0 | 0

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, up to approximately 8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Young TIL | ECCE Young TIL
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, up to approximately 8 months.
Arm/Group | Standard Young TIL | ECCE Young TIL
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Young TIL (N=1) | ECCE Young TIL (N=1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (1) — fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-07-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT01369875/Prot_SAP_000.pdf
  • Informed Consent Form (2012-07-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT01369875/ICF_001.pdf